CLINICAL TRIAL: NCT01171677
Title: Impact of Exercise and Affirmations (IntenSati) on Addiction-related Cognitive and Psychosocial Deficits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: New York University (Other)
Responsible Party: Principal Investigator, John Rotrosen, Professor, NYU Langone Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NYULMC - 10-01156
Record Dates: First submitted 2010-07-27; First posted 2010-07-28 (Estimated); Results first posted 2013-03-06 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-01

CONDITIONS: Drug Dependence; Alcohol Dependence
Keywords: addiction; exercise; cognitive function; mood; self efficacy
MeSH Terms: conditions — Substance-Related Disorders; Alcoholism; Behavior, Addictive; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IntenSati (Experimental): IntenSati (a blending of the words "intention" and "sati," the Pali term for "mindfulness") combines simple yet vigorous physical movements taken from yoga, martial arts, kickboxing and dance with spoken positive affirmation (e.g. "I believe I will succeed", "I am strong" and "I am confident") that are recited simultaneously with the execution of the movements. Indeed, one of the most common reports of IntenSati practitioners is the power of the spoken affirmations to "stick in your head" long after the workout is complete. The literature suggests that both the kind of high level aerobic exercise provided by IntenSati as well as the positive affirmations may have measurable beneficial effects on cognitive function, mood, self efficacy and self esteem.
  Interventions: Behavioral: IntenSati
- Treatment as Usual (No Intervention)

INTERVENTIONS:
Behavioral: IntenSati — IntenSati (a blending of the words "intention" and "sati," the Pali term for "mindfulness") combines simple yet vigorous physical movements taken from yoga, martial arts, kickboxing and dance with spoken positive affirmation (e.g. "I believe I will succeed", "I am strong" and "I am confident") that are recited simultaneously with the execution of the movements. Indeed, one of the most common reports of IntenSati practitioners is the power of the spoken affirmations to "stick in your head" long after the workout is complete. The literature suggests that both the kind of high level aerobic exercise provided by IntenSati as well as the positive affirmations may have measurable beneficial effects on cognitive function, mood, self efficacy and self esteem.
  Other Names: exercise; aerobics; verbal affirmations
  Arms: IntenSati

SUMMARY:
Addiction to illicit and prescribed drugs, alcohol and tobacco is associated with a panoply of brain changes that contribute to structural and micro-structural deficits, altered metabolism and neurotransmission, and related cognitive deficits affecting executive function, decision-making, reward salience and motivation. Many of these deficits may act as barriers to recovery, compromising the same spectrum of cognitive processes that established interventions (motivational enhancement, cognitive behavioral therapy, therapeutic communities, etc.) depend on for successful outcomes. Even where there are medications that target a specific addiction (e.g., methadone for opiates), meaningful, sustained recovery relies on the acquisition of adaptive skills and strategies. As such, there is a need to develop interventions for substance use disorders that have the potential to improve health and cognitive and psychosocial functioning, and to be embraced by the treatment community. A growing body of basic and clinical research suggests that physical exercise may reduce drug use and improve cognitive-executive function, mood, and motivation. There is also a growing literature on the effectiveness of positive affirmation as a cognitive-behavioral intervention for depression and PTSD both of which frequently co-occur with addiction. Building on this, we hypothesize that a combined exercise and affirmation intervention (IntenSati) will lead to improved cognitive and psychosocial function. To test this, we propose to conduct a two-arm randomized clinical trial - in adult volunteers with a history of longstanding substance use and who are in treatment in a residential therapeutic community setting (Odyssey House) - to examine cognitive and psychosocial function before, during, and after randomization to either a twelve-week IntenSati intervention condition or to a twelve-week no-exercise/no-affirmations control condition. This is a pilot study intended to collect data on feasibility and effect size. The population and sample size were selected on the basis of likelihood to benefit from the intervention, likelihood for good adherence, and the realities of completing a low-cost pilot study within a one-year timeframe. Overall there were no substantial differences between IntenSati and TAU on measures of cognition, mood, and psychosocial functioning. Limitations include the small sample size, limited exercise intensity and capacity, missed exercise classes, dropout because of placement, work schedules and non-study-related medical conditions.

DETAILED DESCRIPTION:
Addiction to illicit and prescribed drugs, alcohol and tobacco is associated with a panoply of brain changes that contribute to structural and micro-structural deficits, altered metabolism and neurotransmission, and related cognitive deficits affecting executive function, decision-making, reward salience and motivation. Many of these deficits may act as barriers to recovery, compromising the same spectrum of cognitive processes that established interventions (motivational enhancement, cognitive behavioral therapy, therapeutic communities, etc.) depend on for successful outcomes. Even where there are medications that target a specific addiction (e.g., methadone for opiates), meaningful, sustained recovery relies on the acquisition of adaptive skills and strategies. As such, there is a need to develop interventions for substance use disorders that have the potential to improve health and cognitive and psychosocial functioning, and to be embraced by the treatment community. A growing body of basic and clinical research suggests that physical exercise may reduce drug use and improve cognitive-executive function, mood, and motivation. There is also a growing literature on the effectiveness of positive affirmation as a cognitive-behavioral intervention for depression and PTSD both of which frequently co-occur with addiction. Building on this, we hypothesize that a combined exercise and affirmation intervention (IntenSati) will lead to improved cognitive and psychosocial function. To test this, we propose to conduct a two-arm randomized clinical trial - in adult volunteers with a history of longstanding substance use and who are in treatment in a residential therapeutic community setting (Odyssey House) - to examine cognitive and psychosocial function before, during, and after randomization to either a twelve-week IntenSati intervention condition or to a twelve-week no-exercise/no-affirmations control condition. This is a pilot study intended to collect data on feasibility and effect size. The population and sample size were selected on the basis of likelihood to benefit from the intervention, likelihood for good adherence, and the realities of completing a low-cost pilot study within a one-year timeframe. Overall there were no substantial differences between IntenSati and TAU on measures of cognition, mood, and psychosocial functioning. Limitations include the small sample size, limited exercise intensity and capacity, missed exercise classes, dropout because of placement, work schedules and non-study-related medical conditions.

ELIGIBILITY:
Inclusion Criteria:

1. male or female;
2. 55 or older (resident in OH ElderCare program);
3. able to understand and provide a written informed consent, and agree to adhere to both OH and protocol requirements;
4. meets DSM-IV criteria for drug or alcohol dependence within the previous year;
5. at least a 4 year history of drug/alcohol dependence;
6. receives medical clearance by staff physician.

Exclusion Criteria:

1. medical conditions that contra-indicate intensive physical exercise;
2. body mass index (BMI) greater than 35 kg/m2;
3. cardiovascular disease including untreated high blood pressure (>140/90);
4. other factors that in the opinion of the investigators would either jeopardize the safety of the subject and/or the likelihood of study completion, or compromise the validity of the findings.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-07; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Rotrosen, MD, Principal Investigator — NYU School of Medicine; Wendy Suzuki, PhD, Study Director — New York University; Gary Harmon, PhD, Study Director — Odyssey House

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 Subjects consented, 4 discontinued prior to completing screening, 36 completed baseline, 4 were ineligible, 32 were randomized.
Groups:
- Treatment as Usual: Odyssey House delivers a rich array of services which are typically embedded in Enhanced Therapeutic Community (ETC) settings. The ETC incorporates a highly structured, peer-driven social learning model supported by professional medical, psychiatric, vocational and educational services. Clients create a self-directed treatment plan with definable goals and outcomes and participate in structured group and individual counseling sessions with trained professional staff while living onsite for a period of six to twelve months. Clients attend onsite educational classes and/or participate in onsite job training through job-related tasks and functions within the facility. Regular seminars are conducted to teach life skills, including parenting, anger management, and relapse prevention with the goal of eventual successful reintegration into the community.
Period: Overall Study
Arm/Group | IntenSati | Treatment as Usual
Started | 17 | 15
Completed | 11 | 12
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Adverse Event | 1 | 0
Not completed — completed <70% IntenSati classes | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IntenSati | Treatment as Usual | Total
Number analyzed (Participants) | 17 | 15 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 14 | 28
  >=65 years | 3 | 1 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 59 (4.3) | 59 (3.2) | 59 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 14 | 17
  Male | 14 | 1 | 15
Region of Enrollment [Number; unit: participants]
  United States | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Hopkins Verbal Learning Test (HVLT) Total Recall
Description: The Hopkins Verbal Learning Test (HVLT) assesses Verbal learning and memory, immediate recall, delayed recall, and delayed recognition. The HVLT is comprised of three subscales: HVLT Total Recall, HVLT Delayed Recall, and HVLT Delayed Recognition. HVLT Total Recall is the sum of 3 trials in which twelve words are read to and repeated back by subject. The HVLT Total Recall scale ranges from 0-36, the higher score associated with greater verbal learning.
Time Frame: Baseline to end of intervention (week 14)
Population: participants completing each arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IntenSati | Treatment as Usual
Number analyzed (Participants) | 11 | 12
units on a scale
  HVLT Total (baseline) | 17.27 (3.80) | 18.00 (5.15)
  HVLT Total (end of intervention) | 15.27 (3.98) | 17.50 (3.50)

2. Primary Outcome: Hopkins Verbal Learning Test (HVLT) Delayed Recall
Description: Hopkins Verbal Learning Test (HVLT) assesses Verbal learning and memory, immediate recall, delayed recall, and delayed recognition. The HVLT is comprised of three subscales: HVLT Total Recall, HVLT Delayed Recall, and HVLT Delayed Recognition. HVLT Delayed Recall is administered 20-25 minutes after the HVLT Total Recall. The HVLT Delayed Recall scale ranges from 0-12, the higher score associated with greater retention.
Time Frame: Baseline to end of intervention (week 14)
Population: participants completing each arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IntenSati | Treatment as Usual
Number analyzed (Participants) | 11 | 12
units on a scale
  HVLT Delayed (baseline) | 2.82 (1.72) | 5.00 (2.41)
  HVLT Delayed (end of intervention) | 3.91 (1.76) | 3.92 (2.94)

3. Primary Outcome: Hopkins Verbal Learning Test (HVLT) Delayed Recognition
Description: Hopkins Verbal Learning Test (HVLT) assesses Verbal learning and memory, immediate recall, delayed recall, and delayed recognition. The HVLT is comprised of three subscales: HVLT Total Recall, HVLT Delayed Recall, and HVLT Delayed Recognition. HVLT Delayed Recognition is administered immediately after the HVLT Delayed Recall subscale and involves 12 forced choice responses. The HVLT Delayed Recognition scale ranges from 0-24, the higher score associated with greater recognition ability.
Time Frame: Baseline to end of intervention (week 14)
Population: participants completing each arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IntenSati | Treatment as Usual
Number analyzed (Participants) | 11 | 12
units on a scale
  HVLT Delayed Recognition (baseline) | 18.55 (1.29) | 21.33 (3.37)
  HVLT Delayed Recognition (end of intervention) | 20.27 (1.62) | 22.33 (2.43)

4. Primary Outcome: Stroop Word
Description: Stroop Color Word Test assesses cognitive flexibility, resistance to interference from outside stimuli, creativity, psychopathology and cognitive complexity. The Stroop consists of three subscales: Word, Color, and Color-Word. The Stroop Word test is the first subscale administered. The raw score is determined by the number of correct responses within a 90-second period. The scale ranges from 0-100, the higher score the greater the cognitive flexibility.
Time Frame: Baseline to end of intervention (week 14)
Population: participants completing each arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IntenSati | Treatment as Usual
Number analyzed (Participants) | 11 | 12
units on a scale
  Stroop Word (baseline) | 77.36 (18.48) | 80.67 (20.15)
  Stroop Word (end of intervention) | 83.18 (14.66) | 79.25 (20.21)

5. Primary Outcome: Stroop Color
Description: Stroop Color Word Test assesses cognitive flexibility, resistance to interference from outside stimuli, creativity, psychopathology and cognitive complexity. The Stroop consists of three subscales: Word, Color, and Color-Word. The Stroop Color test is the second subscale administered. The raw score is determined by the number of correct responses within a 90-second period. The scale ranges from 0-100, the higher score the greater the cognitive flexibility.
Time Frame: Baseline to end of intervention (week 14)
Population: participants completing each arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IntenSati | Treatment as Usual
Number analyzed (Participants) | 11 | 12
units on a scale
  Stroop Color (baseline) | 54.27 (14.19) | 64.33 (16.55)
  Stroop Color (end of intervention) | 58.18 (14.74) | 65.67 (15.51)

6. Primary Outcome: Stroop Color/Word
Description: Stroop Color Word Test assesses cognitive flexibility, resistance to interference from outside stimuli, creativity, psychopathology and cognitive complexity. The Stroop consists of three subscales: Word, Color, and Color-Word. The Stroop Color-Word test is the third subscale administered. The raw score is determined by the number of correct responses within a 90-second period. The scale ranges from 0-100, the higher score the greater the cognitive flexibility and resistance to interference.
Time Frame: Baseline to end of intervention (week 14)
Population: participants completing each arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IntenSati | Treatment as Usual
Number analyzed (Participants) | 11 | 12
units on a scale
  Stroop Color/Word (baseline) | 28.82 (9.38) | 33.08 (11.26)
  Stroop Color/Word (end of intervention) | 26.27 (13.79) | 31.17 (11.51)

7. Primary Outcome: Trailmaking Test A
Description: Trailmaking Test A and B measures cognitive shifting, visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning. The test generally requires ability to sequence (Parts A and B), ability to shift cognitive set (Part B), and processing speed (Parts A and B). Part A and Part B are scored separately and expressed in terms of the number of seconds it takes the participant to complete each section, the higher the score the longer it took the subject to complete the test. Trailmaking Part A assesses cognitive processing speed. The lower the score the faster the processing speed.
Time Frame: Baseline to end of intervention (week 14)
Population: participants completing trial
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | IntenSati | Treatment as Usual
Number analyzed (Participants) | 11 | 12
seconds
  Trailmaking A (baseline) | 49.82 (24.15) | 35.99 (12.10)
  Trailmaking A (end of intervention) | 46.98 (21.00) | 38.51 (13.25)

8. Primary Outcome: Trailmaking Test B
Description: Trailmaking Test A and B measures cognitive shifting, visual search speed, scanning, speed of processing, mental flexibility, as well as executive functioning. The test generally requires ability to sequence (Parts A and B), ability to shift cognitive set (Part B), and processing speed (Parts A and B). Part A and Part B are scored separately and expressed in terms of the number of seconds it takes the participant to complete each section, the higher the score the longer it took the subject to complete the test. Trailmaking Part B examines executive functioning and ability to shift cognitive set. The lower the score the faster the ability to shift cognitive set.
Time Frame: Baseline to end of intervention (week 14)
Population: participants completing each arm
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | IntenSati | Treatment as Usual
Number analyzed (Participants) | 11 | 12
seconds
  Trailmaking B (baseline) | 166.07 (66.58) | 126.14 (54.07)
  Trailmaking B (end of intervention) | 187.86 (140.23) | 125.06 (66.27)

9. Primary Outcome: Digit Span
Description: Digit span measures attention efficiency. The Digit-span task is used to measure verbal working memory. Two subscales, Digits Forward and Digits Backward, were combined for a total scale range from 0-30, the higher the score the better the working memory.
Time Frame: Baseline to end of intervention (week 14)
Population: participants completing each arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IntenSati | Treatment as Usual
Number analyzed (Participants) | 11 | 12
units on a scale
  Digit Span (baseline) | 12.55 (2.54) | 12.33 (3.42)
  Digit Span (end of intervention) | 11.91 (3.42) | 12.33 (3.68)

10. Primary Outcome: Controlled Oral Word Association Test (COWAT)
Description: Controlled Oral Word Association Test (COWAT) measures verbal fluency. The assessment consists of three trials; the total score is a sum of all three trials. The scale ranges from 0-90, the higher the score the higher the verbal fluency.
Time Frame: Baseline to end of intervention (week 14)
Population: participants completing each arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IntenSati | Treatment as Usual
Number analyzed (Participants) | 11 | 12
units on a scale
  COWAT (baseline) | 29.91 (10.26) | 31.42 (9.22)
  COWAT (end of intervention) | 27.82 (9.43) | 34.17 (10.70)

11. Primary Outcome: Wechsler Test of Adult Reading (WTAR)
Description: Wechsler Test of Adult Reading (WTAR) measures reading ability. The test involves 50 incorrectly spelled words. The score is computed based on the number of correctly pronounced words. The scale ranges from 0-50, the higher the score the higher the reading ability.
Time Frame: Baseline to end of intervention (week 14)
Population: participants completing each arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IntenSati | Treatment as Usual
Number analyzed (Participants) | 11 | 12
units on a scale
  WTAR (baseline) | 20.73 (9.88) [lower limit 10.92] | 18.17 (10.92)
  WTAR (end of intervention) | 18.18 (9.24) | 17.50 (9.91)

12. Primary Outcome: Self-Efficacy for Abstinence
Description: The Self-Efficacy for Abstinence assessment is adapted from DiClemente (1994)'s Alcohol Abstinence Self-Efficacy. The modified 10-item, 5-point Likert scale (Not at all to Extremely) assesses confidence in abstaining from alcohol. The scale is comprised of four subscales: negative affect, social/positive, physical and other concerns, and withdrawal and urges. Overall abstinence self-efficacy score is calculated by summing each item. The scale ranges from 10-50, the higher the score the higher the self-efficacy for abstinence.
Time Frame: Baseline to end of intervention (week 14)
Population: participants completing each arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IntenSati | Treatment as Usual
Number analyzed (Participants) | 11 | 12
units on a scale
  Self-Efficacy for Abstinence (baseline) | 38.45 (13.19) | 39.58 (9.95)
  Self-Efficacy for Abstinence (end of intervention) | 40.55 (9.53) | 41.17 (10.06)

13. Primary Outcome: Quality of Life (QoL)
Description: The Quality of Life (QoL) assessment is adapted from Quality of Life Enjoyment and Satisfaction Questionnaire (Q-LES-Q). The 23-item QoL consists of five subscales: physical health/activities, feelings, leisure time activities, social relations, and general activities. The scale ranges from 23-115; the higher score indicates higher quality of life enjoyment and satisfaction.
Time Frame: Baseline to end of intervention (week 14)
Population: participants completing intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IntenSati | Treatment as Usual
Number analyzed (Participants) | 11 | 12
units on a scale
  QoL (baseline) | 97.82 (10.00) | 92.17 (10.43)
  QoL (end of intervention) | 92.36 (14.45) | 90.17 (12.83)

14. Primary Outcome: Roesenberg Self Esteem
Description: The Rosenberg Self-Esteem Scale is a 10-item, 4-point Likert scale used to assess global self-esteem. The scale ranges from 0-30 with higher scores indicating higher the self-esteem.
Time Frame: Baseline to end of intervention (week 14)
Population: participants completing each arm
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IntenSati | Treatment as Usual
Number analyzed (Participants) | 11 | 12
units on a scale
  Rosenberg Self-Esteem (baseline) | 23.18 (3.84) | 21.83 (5.01)
  Rosenberg Self-Esteem (end of intervention) | 24.18 (4.31) | 23.33 (4.33)

ADVERSE EVENTS:
Time Frame: Baseline to end of intervention (week 14)
Arm/Group | Intensati | Treatment As Usual
Serious Adverse Events (participants affected / at risk) | 0/17 | 1/15
Other Adverse Events (participants affected / at risk) | 1/17 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensati (N=17) | Treatment As Usual (N=15)
Viral intestinal infection, unspecified (A08.4) (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intensati (N=17) | Treatment As Usual (N=15)
dizziness (R42) and dyspnoea (R06.0) (Cardiac disorders) | 1 (1) | 0 (0) — Occurred prior to initiation of exercise intervention. Subject was excluded from participation in exercise classes.

LIMITATIONS AND CAVEATS:
Overall small sample size, limited exercise intensity and capacity, missed exercise classes, dropout because of placement, work schedules and non-study-related medical conditions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes